CLINICAL TRIAL: NCT00542451
Title: A Phase II Trial of Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Brief Title: Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-199
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Carcinoma of the Breast
Keywords: node-negative breast cancer; HER-2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer (Experimental): 80 mg of paclitaxel per square meter of body-surface area weekly for 12 weeks and a loading dose of 4 mg of intravenous trastuzumab per kilogram of body weight on day 1, followed by 2 mg per kilogram weekly, for a total of 12 doses. After the completion of 12 weeks of treatment with Trastuzumab, the dosing of Trastuzumab could be continued on a weekly basis, or the regimen could be changed to 6 mg per kilogram every 3 weeks for 40 weeks to complete a full year of intravenous treatment with trastuzumab.
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Paclitaxel — Every week for 12 weeks
  Other Names: Taxol
Drug: Trastuzumab — Once a week for twelve weeks Then once a week or once every three weeks for 40 weeks
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to find out what effect the postoperative combination of therapies: trastuzumab (herceptin) and paclitaxel (taxol) will have on breast cancer recurrence. A combination of trastuzuamb and chemotherapy has been used in women with node positive and high risk node negative disease. This tests utilizes a well tolerated regimen of weekly paclitaxel and trastuzumab in women with T1, node negative tumors that are HER2 positive. We would like to determine how effective this drug combination is when used in women with early stage breast cancer, as well as to better define the side effects of this treatment.

DETAILED DESCRIPTION:
* Participants will enroll in this study at the time they are starting their adjuvant therapy for breast cancer. Participants will receive chemotherapy with paclitaxel every week for 12 weeks. They will begin to receive trastuzumab at the same time they begin paclitaxel. Once they have completed the 12 weeks of paclitaxel and trastuzumab, they will receive trastuzumab every 3 weeks or weekly for 40 weeks.
* Participants will be followed with routine assessments such as physical exam and vital signs every 3 months for the first year, and then every 6 months for years 2-5. Then we would like to keep track of the participants medical condition by calling them on the telephone once per year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive carcinoma of the breast
* Tumors must be less than or equal to 3cm in greatest dimension
* Must have node-negative breast cancer according to teh AJCC 7th edition
* ER/PR determination is required. ER- and PR-assays should be performed by immunohistochemical methods
* HER-2 positive: IHC 3+ or FISH >2
* Bilateral breast cancers that individually meet eligibility criteria are allowed
* Patients should have tumor tissue available, and a tissue block of sufficient size to make 15 slides must be sent to DFCI for testing
* Less than or equal to 84 days from mastectomy or from axillary dissection or sentinel node biopsy if the patient's most extensive breast surgery was a breast-sparing procedure
* All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy (lumpectomy), with either a sentinel node biopsy or axillary dissection
* 18 years of age or older
* ECOG Performance Status of 0 or 1
* Adequate bone marrow function, hepatic function, and renal function as outlined in protocol
* Left ventricular ejection fraction of greater than or equal to 50%
* Willingness to discontinue any hormonal agent prior to registration and while on study
* Willingness to discontinue sex hormonal therapy, e.g. birth control pills, prior to registration and while on study
* Patients with a history of ipsilateral DCIS are eligible if they were treated with wide-excision alone, without radiation therapy
* Patients undergoing breast conservation therapy must not have any contraindications to radiation therapy

Exclusion Criteria:

* Pregnant or nursing women
* Locally advanced tumors at diagnosis, including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes
* History of prior chemotherapy in past 5 years
* History of prior trastuzumab therapy
* Active, unresolved infection
* Prior history of any other malignancy in the past 5 years, except for early stage tumors of the skin or cervix treated with curative intent
* Sensitivity to benzyl alcohol
* Grade 2 or greater neuropathy per NCI's CTCAv3.0. (Exception: Any chronic neurologic disorder will be looked at on a case-by-case basis by the study chair).
* Active cardiac disease as outlined in protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2007-10; Primary Completion 2014-04-21 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (20):
- United States (20):
  - University of California-San Francisco, San Francisco, California
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber at Faulkner Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Healthcare, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - North Shore Medical Center, Peabody, Massachusetts
  - Washington University, St Louis, Missouri
  - North Shore LIJ Health System Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Case Western University, Cleveland, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - University of Vermont Cancer Center, Burlington, Vermont

REFERENCES:
- [Derived] Tolaney SM, Tarantino P, Graham N, Tayob N, Pare L, Villacampa G, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis MJ, Shapira I, Wolff AC, Carey LA, Barroso-Sousa R, Villagrasa P, DeMeo M, DiLullo M, Zanudo JGT, Weiss J, Wagle N, Partridge AH, Waks AG, Hudis CA, Krop IE, Burstein HJ, Prat A, Winer EP. Adjuvant paclitaxel and trastuzumab for node-negative, HER2-positive breast cancer: final 10-year analysis of the open-label, single-arm, phase 2 APT trial. Lancet Oncol. 2023 Mar;24(3):273-285. doi: 10.1016/S1470-2045(23)00051-7. PMID 36858723
- [Derived] Tolaney SM, Guo H, Pernas S, Barry WT, Dillon DA, Ritterhouse L, Schneider BP, Shen F, Fuhrman K, Baltay M, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis MJ, Shapira I, Wolff AC, Carey LA, Overmoyer B, Partridge AH, Hudis CA, Krop IE, Burstein HJ, Winer EP. Seven-Year Follow-Up Analysis of Adjuvant Paclitaxel and Trastuzumab Trial for Node-Negative, Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer. J Clin Oncol. 2019 Aug 1;37(22):1868-1875. doi: 10.1200/JCO.19.00066. Epub 2019 Apr 2. PMID 30939096
- [Derived] Barroso-Sousa R, Barry WT, Guo H, Dillon D, Tan YB, Fuhrman K, Osmani W, Getz A, Baltay M, Dang C, Yardley D, Moy B, Marcom PK, Mittendorf EA, Krop IE, Winer EP, Tolaney SM. The immune profile of small HER2-positive breast cancers: a secondary analysis from the APT trial. Ann Oncol. 2019 Apr 1;30(4):575-581. doi: 10.1093/annonc/mdz047. PMID 30753274
- [Derived] Tolaney SM, Barry WT, Dang CT, Yardley DA, Moy B, Marcom PK, Albain KS, Rugo HS, Ellis M, Shapira I, Wolff AC, Carey LA, Overmoyer BA, Partridge AH, Guo H, Hudis CA, Krop IE, Burstein HJ, Winer EP. Adjuvant paclitaxel and trastuzumab for node-negative, HER2-positive breast cancer. N Engl J Med. 2015 Jan 8;372(2):134-41. doi: 10.1056/NEJMoa1406281. PMID 25564897

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer: 80 mg of paclitaxel per square meter of body-surface area weekly for 12 weeks and a loading dose of 4 mg of intravenous trastuzumab per kilogram of body weight on day 1, followed by 2 mg per kilogram weekly, for a total of 12 doses. After the completion of 12 weeks of treatment with Trastuzumab, the dosing of Trastuzumab 6mg/kg over 3 weeks to complete a full year of intravenous treatment with trastuzumab.
Period: Overall Study
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Started | 406
Completed | 327
Not Completed | 79
Not completed — Adverse Event | 31
Not completed — Withdrawal by Subject | 30
Not completed — Physician Decision | 4
Not completed — Recurrent disease | 1
Not completed — unknown reason | 1
Not completed — Death | 2
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Groups:
- Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer: 80 mg of paclitaxel per square meter of body-surface area weekly for 12 weeks and a loading dose of 4 mg of intravenous trastuzumab per kilogram of body weight on day 1, followed by 2 mg per kilogram weekly, for a total of 12 doses. After the completion of 12 weeks of treatment with Trastuzumab.
  Trastuzumab 6mg/kg over 3 weeks to complete a full year of intravenous treatment with trastuzumab.
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 406
Age, Customized [Count of Participants; unit: Participants]
  < 50 yr | 132
  50-59 yr | 137
  60-69 yr | 96
  >= 70 yr | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 351
  More than one race | 0
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: 3-year Disease Free Survival (DFS) Rate
Description: Disease-free survival (DFS) is the proportion of participants ramaing disease free at 3 years based on the Kaplan-Meier method. DFS is defined to end at the time of the first of the following events: local/regional ipsilateral invasive recurrence (or ipsilateral invasive new primary), contralateral invasive breast cancer, distant recurrence, or death from any cause.
Time Frame: at 3 years
Measure: Number (95% Confidence Interval); unit: proportion of participant
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 406
proportion of participant | 0.987 [0.976 to 0.998]

2. Secondary Outcome: Disease Free Survival (DFS) in Patients With Tumors Measuring ≤1 cm or > 1 cm
Description: DFS is defined as the time from registration to the first of the following events: local/regional ipsilateral invasive recurrence (or ipsilateral invasive new primary), contralateral invasive breast cancer, distant recurrence, or death from any cause. Patients without an event are censored at the date of last evaluation.
Time Frame: at 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- [Primary Tumor ≤ 1cm]Adjuvant Paclitaxel + Trastuzumab for Node-Negative HER2-Positive Breast Cancer; [Primary Tumor > 1cm]Adjuvant Paclitaxel + Trastuzumab for Node-Negative HER2-Positive Breast Cancer: 80 mg of paclitaxel per square meter of body-surface area weekly for 12 weeks and a loading dose of 4 mg of intravenous trastuzumab per kilogram of body weight on day 1, followed by 2 mg per kilogram weekly, for a total of 12 doses. After the completion of 12 weeks of treatment with Trastuzumab, the dosing of Trastuzumab could be continued on a weekly basis, or the regimen could be changed to 6 mg per kilogram every 3 weeks for 40 weeks to complete a full year of intravenous treatment with trastuzumab.
Arm/Group | [Primary Tumor ≤ 1cm]Adjuvant Paclitaxel + Trastuzumab for Node-Negative HER2-Positive Breast Cancer | [Primary Tumor > 1cm]Adjuvant Paclitaxel + Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 201 | 205
months | NA [NA to NA] — The lower limit of the 95% confidence interval for the Kaplan Meier curves did not cross 50%. Therefore we cannot get a lower bound of the 95% confidence interval for the median. There are insufficient numbers of participants with events and hence median survival was not reached and the 95% confidence intervals could not be estimated either. | NA [NA to NA] — The lower limit of the 95% confidence interval for the Kaplan Meier curves did not cross 50%. Therefore we cannot get a lower bound of the 95% confidence interval for the median. There are insufficient numbers of participants with events and hence median survival was not reached and the 95% confidence intervals could not be estimated either.

3. Secondary Outcome: Number of Patients With Grade III/IV Cardiac Left Ventricular Dysfunction
Description: cardiac left ventricular dysfunction related adverse events (AE) with any attribution of possibly, probably or definite based on CTCAEv3 as reported on case report forms were counted.
Time Frame: AE evaluated on treatment every week during paclitaxel and every 9 weeks during trastuzumab monotheryapy, and at progression, and observation years 2-10. Median treatment duration was 11.4 months (range 0 - 23.5 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 406
Participants | 2

4. Secondary Outcome: Number of Patients With Grade III/IV Neurotoxicity
Description: Nervous system disorders related adverse events (AE) with any attribution of possibly, probably or definite based on CTCAEv3 as reported on case report forms were counted.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 406
Participants | 13

5. Secondary Outcome: Number of Patients With Amenorrhea
Description: Patients that eligible for amenorrhea assessment and data collecting will be evaluated by standard method defined per protocol 3.9, through menses assessment survey.
Time Frame: Menses Assessment survey on Q6 months x 1 year, then q6months for year 2 and at progression, and observation years 2-10 or until progression.
Population: 64 women are evaluable for the amenorrhea assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
Number analyzed (Participants) | 64
Participants | 18

ADVERSE EVENTS:
Time Frame: AE evaluated on treatment every week during paclitaxel and every 9 weeks during trastuzumab monotheryapy, and at progression, and observation years 2-10. Median treatment duration was 11.4 months (range 0 - 23.5 months).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer
All-Cause Mortality (participants affected / at risk) | 2/406
Serious Adverse Events (participants affected / at risk) | 60/406
Other Adverse Events (participants affected / at risk) | 406/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer (N=406)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Pain (General disorders) | 2
Anaphylaxis (Immune system disorders) | 7
Gum infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 13
White blood cell decreased (Investigations) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9
Irregular menstruation (Reproductive system and breast disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvant Paclitaxel and Trastuzumab for Node-Negative HER2-Positive Breast Cancer (N=406)
Anemia (Blood and lymphatic system disorders) | 20
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 12
Acute coronary syndrome (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 6
Chest pain - cardiac (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2
External ear pain (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1
Flashing lights (Eye disorders) | 2
Watering eyes (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Colonic perforation (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 49
Dyspepsia (Gastrointestinal disorders) | 14
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 8
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 81
Fever (General disorders) | 7
General disorders and administration site conditions - Other, specify (General disorders) | 11
Injection site reaction (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 15
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 28
Immune system disorders - Other, specify (Immune system disorders) | 2
Bladder infection (Infections and infestations) | 4
Bronchial infection (Infections and infestations) | 4
Conjunctivitis infective (Infections and infestations) | 1
Esophageal infection (Infections and infestations) | 2
Gum infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 11
Infective myositis (Infections and infestations) | 2
Nail infection (Infections and infestations) | 2
Phlebitis infective (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Salivary gland infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 9
Skin infection (Infections and infestations) | 17
Soft tissue infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 9
Vaginal infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 6
Burn (Injury, poisoning and procedural complications) | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 6
Fracture (Injury, poisoning and procedural complications) | 2
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 22
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 2
INR increased (Investigations) | 3
Investigations - Other, specify (Investigations) | 4
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 29
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 24
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 29
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Acoustic nerve disorder NOS (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 14
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 48
Sinus pain (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 19
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 22
Proteinuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 4
Urinary tract pain (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Irregular menstruation (Reproductive system and breast disorders) | 8
Pelvic pain (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Uterine pain (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 2
Vaginal inflammation (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 72
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Nail loss (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 14
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 3
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 26
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT00542451/Prot_SAP_000.pdf